CLINICAL TRIAL: NCT03576040
Title: Prognostic Interest of a Whole Body Dynamic PET Acquisition in Pre-therapeutic 68Ga-DOTATOC PET/CT for Neuroendocrine Tumors
Brief Title: Whole Body Dynamic 68Ga-DOTATOC PET/CT in Neuroendocrine Tumors
Acronym: GAPET-NET
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: GAPET-NET (29BRC17.0036)
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Neuroendocrine Tumors
Keywords: Positron Emission Tomography Computed Tomography; whole body dynamic acquisition; Gallium 68
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Whole Body Dynamic 68Ga-DOTATOC PET/CT — 68Ga-DOTATOC PET-CT will be performed in the nuclear medicine department of the University Hospital of Brest on a Biograph mCT S64 machine (Siemens medical, Erlangen, Germany) "Time of Flight" system after intravenous injection of 150MBq of 68Ga-DOTATOC. In the usual conditions for performing this exam, the patient must remain at a strict rest for 60 minutes following the injection of the tracer and before a static 3D acquisition. For this protocol, a complementary 4D dynamic acquisition (15-60 minutes post-injection) will be performed during this usual rest period.

SUMMARY:
Neuroendocrine tumors (NET) are a network of rare tumors with common embryological origin. Functional imaging plays a major role in the extension assessment and tumor characterization of NETs. SPECT/CT with 111In-pentetreotide is the recommended test when tumors are well differentiated (grade G1 or G2). It has a real interest in diagnosis, in therapeutic decision-making (in particular by cold somatostatin analogues or in PRRT) and in the systematic follow-up of patients. Nevertheless, SPECT/CT procedure makes for a relatively long review. In addition, scintigraphy has a lower spatial resolution than PET technology and remains of limited interest for signal quantification.

However, the ability to locate and quantitatively measure the absorption of radiopharmaceuticals in the target tissues is a major challenge in oncology for the characterization of the disease.

Recent developments in radiopharmacy have made it possible to target NETs in PET imaging through the use of somatostatin analogues coupled with positron emitters, called 68Ga-DOTA peptides. The diagnostic performance of 68Ga-DOTApeptide PET/CT appears to be superior to SPECT/CT with 111In-pentetreotide. A marketing authorization has thus recently been issued in France for the use of 68Ga-DOTATOC.

Historically, the recommended quantification method in PET was based on the instantaneous measurement in static acquisition (3D) of the maximum of the standardized uptake value (SUVmax). This approach has the disadvantage to measure the signal at a time "t" for a single voxel of the image. Dynamic acquisition methods (4D) have been proposed to extract a radiotracer absorption coefficient (Ki) for a lesion. Several studies have demonstrated the superiority of Ki versus SUVmax in 18FDG PET/CT for the diagnostic management, therapeutic evaluation and prognosis of various solid cancers.

However, no work has validated this approach in PET / CT at 68Ga-DOTATOC as part of the prognostic evaluation of NETs.

The objective of the study is to evaluate the prognostic value of the tumor absorption coefficient Ki resulting from a 4D whole-body dynamic acquisition in PET / CT at 68Ga-DOTATOC in patients with well-differentiated NETs grade I or II according to the WHO classification

ELIGIBILITY:
Inclusion Criteria:

* Patient majeur ≥ 18 year old
* Présenting a well differentiated neuroendocrine tumor (G1 ou G2)
* Indication performing a68Ga-DOTATOC PET/CT
* non-opposition

Exclusion Criteria:

* Patient <18 years old
* Breastfeeding/ pregnancy
* Other type of tumor
* Refusal of participation

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with NET histologically proven and presented in RCP RENATEN at CHRU Brest Primitive: Gastroenteropancreatic, bronchopulmonary or unknown
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  To evaluate the prognostic value of lesionnal Ki on progression-free survival at 2 years and compare it with SUVmax (static 3D acquisition) in patients with metastatic well-differentiated NET
Recidive free survival (RFS) | 2 years
  To evaluate the prognostic value of Ki lesion on progression-free survival at 2 years and compare it with SUVmax (static 3D acquisition) in patients with localised well-differentiated NET

SECONDARY OUTCOMES:
Correlation between lesionnal Ki and immunochemistry markers | 0 to 2 years
  Evaluate the statistical correlation between lesional Ki versus SUVmax with NET immunohistochemistry markers expression (SSTR2, SSTR3, and SSTR5; BCL2, Phospho-MTOR expression PD-L1 by tumor cells and immune cells, intra-tumor CD8 + lymphocytes, tumor necrosis surface)
Predictive value of non-event survival (PFS+RFS) | 6 months to 2 years
  To evaluate the predictive value of non-event survival (PFS+RFS) with a ΔKi approach in patients receiving an intermediate therapeutic assessment examination (somatostatin analogues or PRRT with 177Lu-DOTATATE), and compare it with a ΔSUVmax approach
Correlation between 68Ga-DOTATOC PET/CT and/or 111In-pentetréotide SPECT/CT and 177Lu-DOTATATE SPECT/CT | 0 to 2 years
  Evaluate the statistical correlation between the SUVmax assessed with 68Ga-DOTATOC PET/CT and/or 111In-pentetréotide SPECT/CT and 177Lu-DOTATATE SPECT/CT
Prognostic value of Ki versus usual prognostic parameters | 2 years
  To evaluate the prognostic value on non-event survival (PFS+RFS) at 2 years of Ki and clinical parameters (sex, age), biological (CgA assay), pathology (grade, differentiation, Ki67 expression, BCL2, phospho-MTOR).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement